CLINICAL TRIAL: NCT06448013
Title: A Phase I Study Investigating the Combination of the Menin Inhibitor Ziftomenib With Venetoclax and Gemtuzumab in Pediatric Patients With Acute Myeloid Leukemia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Kura Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-0911; NCI-2024-04821 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2024-06-03; First posted 2024-06-07 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — venetoclax; Gemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dose Escalation + Dose Expansion (Experimental): Participants found to be eligible to take part in this study, you will be assigned to a dose level of ziftomenib based on when you join this study. Up to 4 dose levels of ziftomenib will be tested. Up to 6 participants will be enrolled at each dose level. The first group of participants will receive the lowest dose level. Each new group will receive a higher dose than the group before it, if no intolerable side effects were seen. This will continue until the recommended dose of ziftomenib is found.
  Interventions: Drug: Venetoclax; Drug: Gemtuzumab; Drug: Ziftomenib

INTERVENTIONS:
Drug: Venetoclax — Given by PO
  Other Names: ABT-199; GDC-0199
Drug: Gemtuzumab — Given by IV
  Other Names: Gemtuzumab ozogamicin; Mylotarg
Drug: Ziftomenib — Given by PO

SUMMARY:
To find the recommended dose of ziftomenib in combination with gemtuzumab ozogamicin and venetoclax that can be given to pediatric participants who have relapsed or refractory AML or MPAL.

DETAILED DESCRIPTION:
Primary Objectives:

- To determine the safety, tolerability, and recommended Phase II dose (RP2D) of ziftomenib in combination with gemtuzumab ozogamicin and venetoclax for pediatric participants with acute myeloid leukemia (AML).

Secondary Objectives:

* To determine the preliminary assessment of efficacy by overall response (OR), including complete remission (CR), CR with incomplete blood count recovery and partial remission, overall survival (OS), event-free survival (EFS) and duration of response (DOR) of pediatric participants treated with this combination.
* To determine time to first response and time to best response of pediatric participants treated with this combination.

Exploratory Objective

- To evaluate molecular and cellular markers that may be predictive of antitumor activity and/or resistance.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 3 year to 21 years
2. Karnofsky for children >16yo and Lansky <16yo.
3. Relapsed/refractory AML, or MPAL with a myeloid phenotype.

   1. Evidence of leukemia (AML, MPAL with a myeloid phenotype) in the bone marrow as detected by morphology or molecular diagnostics.
   2. Presence of KMT2Ar, NUP98r, NPM1c, UBTF-ITD or other HOX pathway mutation.
4. WBC must be below 25,000/ƒÊL at time of enrollment. Participants may receive cytoreduction prior to enrollment.
5. Baseline ejection fraction must be > 40%.
6. Adequate hepatic function (direct bilirubin < 1.5x upper limit of normal (ULN) unless increase is due to Gilbert's disease or leukemic involvement, and AST and/or ALT < 3x ULN unless considered due to leukemic involvement, in which case direct bilirubin or AST and/or ALT < 5x ULN will be considered eligible).
7. Adequate renal function (creatinine clearance ≥ 30 mL/min) unless related to disease.
8. In the absence of rapidly proliferative disease, the interval from prior treatment to time of initiation will be at least 14 days for cytotoxic or non-cytotoxic (immunotherapy agent(s), or an interval of 5 half-lives of the prior therapy. Oral hydroxyurea and/or cytarabine (up to 2 g/m2) for participants with rapidly proliferative disease is allowed before the start of study therapy, as needed, for clinical benefit and after discussion with the PI. Concurrent therapy for central nervous system (CNS) prophylaxis or continuation of therapy for controlled CNS disease is permitted.
9. 3 month washout prior from bone marrow transplantation.
10. Unless surgically or biologically sterile: Women of childbearing potential must agree to adequate methods of contraception during the study and at least 3 months for males, and 6 months for females, after the last treatment.

Exclusion Criteria:

1. Participants who weigh less than 10kg.
2. Participants with any concurrent uncontrolled medical condition, laboratory abnormality, or psychiatric illness which could place the patient at unacceptable risk of study treatment.
3. The use of other chemotherapeutic agents or anti-leukemic agents is not permitted during study with the following exceptions (1) intrathecal chemotherapy for prophylactic use or for controlled CNS leukemia. (2) use of hydroxyurea for patients with rapidly proliferative disease or for control of counts during differentiation syndrome. (3) use of steroids for treatment of differentiation syndrome.
4. Participants with any severe gastrointestinal or metabolic condition which could interfere with the absorption of oral study medications.
5. Participants with chronic liver disease.
6. Participants with a concurrent active malignancy under treatment.
7. Known active hepatitis B (HBV) or Hepatitis C (HCV) infection or known HIV infection.
8. Female participants who are pregnant or breast-feeding.
9. Participants has an active uncontrolled infection.
10. Any of the following within the 6 months prior to study entry: myocardial infarction, uncontrolled/unstable angina, congestive heart failure (New York Heart Association Classification Class ≥II), life-threatening, uncontrolled arrhythmia, cerebrovascular accident, or transient ischemic attack.
11. Mean corrected QT interval by Fredericia's formula >480 ms on triplicate 12-lead electrocardiograms performed within approximately 5 minutes of each other.
12. History of or any concurrent condition, therapy, or laboratory abnormality that in the Investigator's opinion might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the patient to participate.
13. Clinically active central nervous system (CNS) leukemia.
14. The use of topical steroids for cutaneous graft-versus-host disease (GVHD) or stable systemic steroid doses less than or equal to 20 mg of prednisone daily are permitted.
15. Participants with Grade > 2 active acute GVHD, moderate or severe limited chronic GVHD, or extensive chronic GVHD of any severity.

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Estimated)
Dates: Start 2025-03-07 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Branko Cuglievan, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org